CLINICAL TRIAL: NCT06263400
Title: The Effect Of Caregiver Psychoeducation On Recovery Levels Of Depression Patients And Family Burden And Expression Of Emotions Of Caregivers
Brief Title: Recovery Levels of Depression Patients and Caregiver Psychoeducation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Serife Oztaban, principal investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: randomized trial
Record Dates: First submitted 2024-01-14; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Psychoeducation
Keywords: depressive disorders; Family Burden; Emotional Expression; Psychoeducation
MeSH Terms: conditions — Depressive Disorder | interventions — Follow-Up Studies

STUDY DESIGN:
Intervention Model Description: In randomization, among the patients who volunteered to participate in the study, the odd number of patients and their caregivers in the list made according to the order of hospitalization constituted the study group, and the even number of patients and their caregivers formed the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation (Experimental): Experimental:Experimental group ın the first meeting with the patients and their caregivers in the experimental group, information about the training was given, information about the patient was obtained, and training days were determined.Structured education and follow-up In the study, we hypothesized that the caregiver psychoeducation program (consisting of six sessions over a 3-week period) would improve depressive symptoms in depressed patients, increase recovery levels, reduce the caregiver's burden, and reduce emotional expression levels in the family.Structured education and follow-up In the study, we hypothesized that the caregiver psychoeducation program (consisting of six sessions over a 3-week period) would improve depressive symptoms in depressed patients, increase recovery levels, reduce the caregiver's burden, and reduce emotional expression levels in the family.
  Interventions: Behavioral: psychoeducation and follow-up study
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Behavioral: psychoeducation and follow-up study — In the study, we hypothesized that the caregiver psychoeducation program (consisting of six sessions over a 3-week period) would improve depressive symptoms in depressed patients, increase recovery levels, reduce the caregiver's burden, and reduce emotional expression levels in the family.
  Arms: Psychoeducation

SUMMARY:
To determine the effect of psychoeducation given to patients and caregivers on patients' depression and recovery levels, caregivers' emotional expression and family burden levels.

DETAILED DESCRIPTION:
The samples of the research are 'The experiment that was followed up in the inpatient service at Adnan Menderes University Research and Practice Hospital Psychiatry Service with diagnoses of F32 (Depressive Disorder according to ICD 10 code) and F33 (Recurrent Depressive Disorder according to ICD 10 code) and met the inclusion criteria for the study (n = 46). ) and a control group (n=46) with a total of 92 depression patients and their caregivers. The experimental group patients and their caregivers and their relatives were included in the psychoeducation program application within the framework of the training recommended in the "Guide for the Treatment of Patients with Major Depressive Disorder" published by APA in 2010. This application is a psychosocial treatment program consisting of structured sessions and including an experiential interactional process. Data were collected from patients using the Beck Depression Scale, Recovery Assessment Scale; It was collected by caregivers using the Emotional Expression Scale and Zarit Family Burden Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection criteria included in the sample for the research;
* Being 18 years or older
* Receiving inpatient treatment with a diagnosis of F32 (Depressive Disorder) or F33 (Recurrent Depressive Disorder)
* Does not have a developmental disorder
* Without psychotic features
* Not having communication problems
* Being at least a primary school graduate Caregiver selection criteria included in the sample for the research;
* Being 18 years or older
* Being the primary caregiver of the patient
* Being at least a primary school graduate

Exclusion Criteria:

* • Patient selection criteria for exclusion from the sample for the research;

  * DSM-V Axis I comorbidity Caregiver selection criteria for exclusion from the sample for the research;
  * With mental retardation or psychotic disorder
  * Having speech and hearing disorders
  * It was created as having one of the diagnoses of a cognitive disorder such as delirium, dementia, or amnestic syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
to patients before training | 1 week after admission
  Depressive symptoms of the patients will be evaluated with the 'Beck Depression Scale'. The scale was developed in 1961, and its Turkish validity and reliability study was conducted in 1989. The scale, which includes the physical, emotional, cognitive and motivational symptoms seen in depression, aims to objectively determine the degree of depression symptoms. It is stated that as the score obtained from the scale increases, the severity of depression also increases. The subjective recovery processes of the patients will be evaluated with the 'recovery evaluation scale'. Turkish validity and reliability study was conducted in 2017. The scale is a 24-item, 5-point Likert type scale. A high total score obtained from the scale indicates that the improvement is high.
pre-training caregivers | 1 week after admission
  The 'healing evaluation scale', a scale consisting of 41 items that determines the emotional expression style and level of patient relatives, was developed in 1993. As the scores increase on the scale, which is answered as "True (1)-False (0)" and is rated between 0-1, the level of emotional expression increases. High scores from the scale are interpreted as a high level of negative reflection of the caregiver's emotional expression, and low scores mean a low level of negative reflection of the caregiver's emotional expression. 'Zarit family burden scale' was developed in 1980, and the Turkish validity and reliability study of the scale was conducted in 2009. The scale consists of 22 statements and is a 5-point Likert type scale. High scores from the scale are interpreted as a high burden level of the caregiver, and low scores mean a low burden level.

SECONDARY OUTCOMES:
after training | 1 month after training
  The Beck depression scale will be used to determine the degree of depression symptoms. The recovery assessment scale will be used to evaluate the subjective recovery processes of depression patients.
  Emotional expression scale will be used to determine caregivers' emotional expression style and level. Zarit family burden scale will be used to measure the burden level of caregivers.
after training | 3 months after training
  The Beck depression scale will be used to determine the degree of depression symptoms. The recovery assessment scale will be used to evaluate the subjective recovery processes of depression patients.
  Emotional expression scale will be used to determine caregivers' emotional expression style and level. Zarit family burden scale will be used to measure the burden level of caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Şerife ÖZTABAN, MsC, Study Chair — AydınAdnan Menderes University, Faculy of Nursing, Division Public Health Nursing
Locations (1):
- AydınAdnan Menderes University, Faculy of Nursing, Division Public Health Nursing, Aydin, Aydın/Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.